CLINICAL TRIAL: NCT05613335
Title: Minimal Invasive Crestal Sinus Technique Using Autologous Fibrin Glue Versus Sticky Bone With Simultaneous Implant Insertion. A Prospective Study
Brief Title: Crestal Sinus Technique Using Autologous Fibrin Glue Vs Sticky Bone With Simultaneous Implant Insertion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M02150620
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Missed Upper Posterior Teeth
Keywords: Crestal sinus lift; Autologous fibrin glue; Sticky bone
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fibrin glue group (Experimental): Maxillary sinus augmentation using autologous fibrin glue with simultaneous implant placement
  Interventions: Procedure: Maxillary sinus augmentation using autologous fibrin glue with simultaneous implant placement
- sticky bone group (Experimental): Maxillary sinus augmentation using mixture of autologous fibrin glue with bone graft with simultaneous implant placement
  Interventions: Procedure: Maxillary sinus augmentation using mixture of autologous fibrin glue with bone graft with simultaneous implant placement

INTERVENTIONS:
Procedure: Maxillary sinus augmentation using autologous fibrin glue with simultaneous implant placement — Maxillary sinus augmentation using autologous fibrin glue with simultaneous implant placement
  Arms: fibrin glue group
Procedure: Maxillary sinus augmentation using mixture of autologous fibrin glue with bone graft with simultaneous implant placement — Maxillary sinus augmentation using mixture of autologous fibrin glue with bone graft with simultaneous implant placement
  Arms: sticky bone group

SUMMARY:
prospective comparison of minimal Invasive Crestal Sinus Technique Using Autologous Fibrin Glue Vs Sticky Bone with simultaneous implant insertion.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical and radiographic outcomes of applying fibrin glue versus sticky bone in conjunction with crestal sinus lift technique associated with simultaneous implant insertion.

ELIGIBILITY:
Inclusion Criteria:

- a) Patients should be willing to be present for regular timely follow up. b) Residual bone height range from 5 to 9mm c) Patent ostium of maxillary sinus. d) Patients having missing maxillary posterior teeth. e) Patient cooperation and compliance are indispensible for a predictable clinical outcome.

f) Patients free from any systemic disease

Exclusion Criteria:

* 1) Patients with systemic disease that prevent surgical intervention or bone healing.

  2) Patients with acute or chronic maxillary sinusitis. 3) Patients with cyst, tumor or root tips at the planned surgical site. 4) Heavy smoker patients. 5) Elderly patients (over 60 years). 6) Patients with Poor oral hygiene or aggressive periodontal diseases. 7) Lack of motivation or inability to maintain oral hygiene.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-18 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 3 months
  implant stability using The Ostell ISQ scale: The ISQ scale ranges from 0 to 100 that measures implant stability. The values less than 60 indicate low implant stability; values from 60 to 69 indicate medium stability where values between 70 and 79 indicate high stability.
  6 implants from each group will be assessed regarding implant stability at 3 months post-operative using this ISQ scale to determine implant stability and data will be analyzed statistically for significance.
Bleeding | 3 months
  Peri-implant mucosal bleeding will be graded using criteria of modified sulcus bleeding index (mBI).
  * Score 0; no bleeding when a periodontal probe was passed along the gingival margin adjacent to the implant.
  * Score 1; isolated bleeding visible spot.
  * Score 2; a confluent red line on the gingival margin was formed by blood.
  * Score 3; heavy or profuse bleeding is present.
Radiographic evaluation | immediate postoperative
  Cone beam computed tomography scan will be taken at preoperative visit to assess:Residual bone height (RBH) which is the distance from the alveolar crest to the floor of the maxillary sinus at the intended implant placement site.
  * Implant protrusion (IP):measured as the distance from the sinus floor to implant apex.
  * Graft height apically (GHa):the distance fom implant apex to the highest level of the grafting material (the new sinus floor).
  * Grafted sinus height (GSH):the distance from the original sinus floor to the new sinus floor which is the implant protrusion plus the graft height beyond the implant apex (IP +GHa).

SECONDARY OUTCOMES:
implant stability | 6 months
  implant stability using The Ostell ISQ scale: The ISQ scale ranges from 0 to 100 that measures implant stability. The values less than 60 indicate low implant stability; values from 60 to 69 indicate medium stability where values between 70 and 79 indicate high stability.
  6 implants from each group will be assessed regarding implant stability at 3 months post-operative using this ISQ scale to determine implant stability and data will be analyzed statistically for significance.
Bleeding | 6 months
  Peri-implant mucosal bleeding will be graded using criteria of modified sulcus bleeding index (mBI).
Radiographic evaluation | 6 months
  Cone beam computed tomography scan will be taken at preoperative visit to assess:Residual bone height (RBH) which is the distance from the alveolar crest to the floor of the maxillary sinus at the intended implant placement site.
  * Implant protrusion (IP):measured as the distance from the sinus floor to implant apex.
  * Graft height apically (GHa):the distance fom implant apex to the highest level of the grafting material (the new sinus floor).
  * Grafted sinus height (GSH):the distance from the original sinus floor to the new sinus floor which is the implant protrusion plus the graft height beyond the implant apex (IP +GHa).

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: No